CLINICAL TRIAL: NCT01198912
Title: Influence of Oral Doxycycline on Wound Healing After Endonasal Endoscopic Sinus Surgery for Chronic Rhinosinusitis With and Without Nasal Polyposis: a Double-blind Randomized Placebo-controlled Trial.
Acronym: DOXYPOSTOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010/384
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Chronic Rhinosinusitis; Nasal Polyps
Keywords: rhinosinusitis; doxycycline; Chronic rhinosinusitis with or without nasal polyps
MeSH Terms: conditions — Nasal Polyps; Rhinosinusitis | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- doxycycline 100 mg (Experimental)
  Interventions: Drug: doxycycline 100 mg

INTERVENTIONS:
Drug: placebo — during 56 days
  Arms: placebo
Drug: doxycycline 100 mg — during 56 days
  Arms: doxycycline 100 mg

SUMMARY:
This is a randomized, double blind, placebo controlled, parallel group, study in patients with chronic rhinosinusitis with or without nasal polyps. The objective is to test the clinical efficacy of long-term low dose oral doxycycline on wound healing quality after endoscopic sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age, of either sex and any race
* diagnosis of chronic rhinosinusitis with or without nasal polyposis according to the EPOS guidelines research
* Subjects should be regularly scheduled for bilateral functional endonasal endoscopic sinus surgery
* Subjects must be in good health, free of any clinically significant disease that would interfere with the study schedule or procedures or compromise his/her safety.
* Subjects must be willing to give informed consent and adhere to visit schedules, medication restrictions, and agree to perform daily diary entries.
* Nonpregnant women of childbearing potential must use a medically acceptable, adequate form of birth control.

Exclusion Criteria:

* Women must not be pregnant, breast feeding, or premenarcheal.
* Subjects who have required oral corticosteroids within the previous four weeks prior to surgery.
* Subjects who have required nasal corticosteroids within the previous one week prior to surgery.
* Subjects with known allergic reaction on tetracyclines, diabetes (type 1 and 2), renal insufficiency, severe liver disease, systemic diseases affecting the nose (e.g. M. Wegener), prior surgeries of the paranasal sinuses.
* Patients with the following diseases should be excluded :

  1. Cystic fibrosis based on positive sweat test or DNA alleles
  2. Gross immunodeficiency (congenital or acquired)
  3. congenital mucociliary problems e.g. primary ciliary dyskinesia (PCD)
  4. Non-invasive fungal balls and invasive fungal disease
  5. systemic vasculitis and granulomatous diseases
  6. Cocaine abuse
  7. Neoplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-11-22 (Actual); Primary Completion 2016-09-06 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
Endoscopic evaluation of quality and speed of wound healing | at 3 months after first drug intake
Recurrence of nasal polyps | at 3 months after first drug intake
Recurrence of nasal polyps | at 6 months after first drug intake

SECONDARY OUTCOMES:
nasal and exhaled NO | at 3 months after first drug intake
nasal and exhaled NO | at 6 months after first drug intake
subjective assessment of the wound healing | at 3 months after first drug intake
subjective assessment of the wound healing | at 6 months after first drug intake
chronic rhinosinusitis symptoms by the patients | at 3 months after first drug intake
chronic rhinosinusitis symptoms by the patients | at 6 months after first drug intake
Questionnaires: SNOT 22, RSOM, SF36 asthma control questionnaire | at 3 months after first drug intake
Questionnaires: SNOT 22, RSOM, SF36 asthma control questionnaire | at 6 months after first drug intake
inflammatory mediators in nasal fluid as well as in serum | at 3 months after first drug intake
inflammatory mediators in nasal fluid as well as in serum | at 6 months after first drug intake

CONTACTS AND LOCATIONS:
Overall Officials: Claus Bachert, MD, PhD, Principal Investigator — University Hospital Ghent, Belgium
Locations (2):
- University Hospital Ghent, Ghent, Belgium
- Univ.-HNO-Klinik, St. Elisabeth Hospital, Bochum, Germany

REFERENCES:
- See also: website University Hospital Ghent, Belgium — http://www.uzgent.be